CLINICAL TRIAL: NCT03353168
Title: Childbirth Related Fear and Worry During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mid Sweden University (Other)
Collaborators: Örebro University, Sweden (Other); Jämtland County Council, Sweden (Other Government); Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/372-31Ö
Record Dates: First submitted 2017-07-19; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Fear of Childbirth; Anxiety
Keywords: fear; anxiety; childbirth; pregnancy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study of childbirth related anxiety, fear or worry, in which we follow women from mid pregnancy until about 8 months postpartum. Our overall aim is to enhance our understanding of psychological factors contributing to childbirth related fear or worry. Specifically, we wish to investigate

* associations between psychological factors (pain catastrophizing, intolerance of uncertainty, worry beliefs, cognitive avoidance, insomnia, life satisfaction, anxiety- and depressive symptoms, worry parameters, and behavioral avoidance) and childbirth related fear or anxiety during pregnancy
* the impact of childbirth related fear or anxiety and other psychological factors during pregnancy on epidural use during delivery and obstetric outcome variables
* childbirth related fear or anxiety during pregnancy, psychological factors, epidural use, and obstetric outcome variables as predictors of self-reported birth experiences 6-10 months postpartum.
* childbirth related fear or anxiety during pregnancy, psychological factors, epidural use, obstetric outcome variables, and self-reported birth experiences as predictors of childbirth related fear or anxiety 6-10 months postpartum

Women in mid-pregnancy will be recruited at routine check-ups with midwifes working in antenatal health care units in two Swedish regions. After consenting to participate, they will be answering a questionnaire with sociodemographic and obstetric background data, measures of childbirth related fear and anxiety, and measures of psychological variables with a potential relation to childbirth related anxiety. 6-10 months after giving birth they will be contacted again with a postpartum follow-up questionnaire asking questions about the experience of giving birth, postpartum levels of childbirth related fear or anxiety, and thoughts about possible future childbirths. They will also be asked if willing to let the research team include information from their obstetric medical chart (e.g. birth mode and birth interventions, use of analgesia, and complications for the mother and baby) in statistical analyses.

DETAILED DESCRIPTION:
Aim and main research questions:

The overall aim with this study investigate psychological factors contributing to childbirth related fear or worry. Specifically, we wish to investigate

* associations between psychological factors (pain catastrophizing, intolerance of uncertainty, worry beliefs, cognitive avoidance, insomnia, life satisfaction, anxiety- and depressive symptoms, worry parameters, and behavioral avoidance) and childbirth related fear or anxiety during pregnancy
* the impact of childbirth related fear or anxiety and other psychological factors during pregnancy on epidural use during delivery and obstetric outcome variables
* childbirth related fear or anxiety during pregnancy, psychological factors, epidural use, and obstetric outcome variables as predictors of self-reported birth experiences 6-10 months postpartum.
* childbirth related fear or anxiety during pregnancy, psychological factors, epidural use, obstetric outcome variables, and self-reported birth experiences as predictors of childbirth related fear or anxiety 6-10 months postpartum

Procedure:

Pregnant women will be recruited by midwives working in antenatal health care units in two Swedish regions; Jämtland/Härjedalen and Örebro County. Recruitment is planned to take place during the first visit following the routine ultrasound examination (normally provided in gestational week 16-20). Women found not eligible will be counted by each antenatal midwife and reported to the project group without any personal identification. Before invited to participate, eligible women will be given oral and written information about the study. Any questions might be asked the midwife directly or via telephone or e-mail to the members of the research group. If accepting participation, each woman will give her written consent. The woman will then receive the first questionnaire. The questionnaire is coded with a unique code for each participant, and does not include any personal identification. It is returned to the research group in a pre-paid envelope. The consent form, also including the unique code of each participant, contact information and personal identification number, is collected by the midwife and later sent to the research group.

In phase two of the study, data will be gathered from two different sources - (a) from the medical birth records of the particular birth, and (b) via a postpartum follow-up questionnaire. These data will be gathered 6-10 months after the planned date of the birth. All women who have returned the first questionnaire and whose address can be confirmed will be contacted by mail and invited to participate in phase two. Letters will be sent, including information about phase two of the project, a postpartum follow-up questionnaire, and a consent form in which the woman can give her written consent for the research team to extract data from the medical birth record. The women are thus free to choose their participation in the two parts of phase 2 separately. The follow-up questionnaire and consent form will returned to the research group by mail, in a pre-paid envelope.

Extraction of medical data: Once consent has been received, obstetric data will be extracted from the medical chart, with help from a midwife at each hospital. The data will be anonymized before leaving the hospital, erasing all personal data such as name and personal identification number, coding the obstetric set of data with the unique participant code number of each woman.

Data and measurements:

The first questionnaire, in mid-pregnancy includes the following sections and scales:

* Sociodemographic background (age, civil status, educational level, occupational status, country of birth)
* Obstetric history/background (pregnancy week, number of fetuses, current pregnancy complications, previous births including birth mode and year)
* Negative experiences in health care
* Preferred mode of birth
* the Fear of Birth Scale, FOBS
* the Wijma Delivery Expectancy/Experience Questionnaire, W-DEQ A
* the Hospital Anxiety and Depression Scale, HADS
* the Pain Catastrophizing Scale, PCS
* the Intolerance of Uncertainty Inventory, part B
* Why Worry II
* the Cognitive Avoidance Questionnaire
* the Insomnia Severity Index, ISI
* the Satisfaction With Life Scale, SWLS
* the Situational Fear of Childbirth, SFC
* items regarding worry frequency, controllability and excess from the GAD-7
* items regarding childbirth specific behavioral avoidance

The postpartum follow-up questionnaire includes:

* Birth information (birth date, birth mode including indication, usage of epidural analgesia)
* the Wijma Delivery Expectancy/Experience Questionnaire, W-DEQ A
* the Fear of Birth Scale, FOBS
* The Childbirth Experience Questionnaire
* Two visual analogue scales regarding the experience of giving birth (vaginally or with Caesarean section) using the anchors "not at all positive" to "very positive" and "not at all negative" to "very negative".
* One visual analogue scale regarding the worst experience of pain during birth, using the anchors "not painful at all" and "worst pain possible".
* One visual analogue scale regarding overall experience of pain during birth, again using the anchors "not painful at all" and "worst pain possible".
* Preferred mode of birth in a future birth

Medical birth data that will be extracted:

* Age of the mother, parity, and gestational week
* Comorbidity
* Obstetric and neonatal outcome variables (see outcome measures)

ELIGIBILITY:
Inclusion Criteria:

* Gestational week 16 or more
* Normal routine ultrasound examination
* Mastery of Swedish language (being able to understand study information and questionnaires)

Exclusion Criteria:

* For extraction of medical birth records: giving birth in another Swedish region than Jämtland/Härjedalen or Örebro county, or giving birth in another country.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A general sample of pregnant Swedish women, recruted at antenatal health care units within primary care.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Birth Scale | Baseline (around gestational week 20-25) and 6-12 months after expected delivery
  Two item VAS-scale assessing worry and fear relating to childbirth. The instrument will be used both as a continuous measure of level of fear, and with a cut point of ≥ 60 indicating fear of birth (< 60 = no fear of birth)
Wijma Delivery Expectancy/Experience Questionnaire | Baseline (around gestational week 20-25) and 6-12 months after expected delivery
  33 item 6 point Likert scale questionnaire in which the items refer to cognitive and emotional expectations of the forthcoming childbirth. The instrument will be used both as a continuous measure of level of fear, and with a cut point of ≥ 85 indicating fear of childbirth (< 85 = no fear of childbirth)

SECONDARY OUTCOMES:
The use of epidural anesthesia during delivery | during delivery
  Use of epidural anesthesia (yes/no) during delivery as reported in obstetric medical chart
Start of contractions | during delivery
  Induced or spontaneous start of contractions
Use of analgesics | during delivery
  Use of analgesics other than epidural
Mode of delivery | during delivery
  Vacuum extraction, forceps, Caesarean or vaginal delivery
Blood loss | during delivery
  Blood loss
APGAR score | after delivery
  APGAR at 1, 5 and 10 minutes
Birth weight | after delivery
  Birth weight
Admission to neonatal ward | after delivery, within 24 hours
  Admission to neonatal ward
Preferred mode of birth | Baseline (around gestational week 20-25) and 6-12 months after expected delivery
  Preferred mode of birth (vaginal or Caesarean)
Experience of giving birth | 6-12 months after expected delivery
  Two 100 mm visual analogue scales regarding the experience of giving birth (vaginally or with Caesarean section) using the anchors "not at all positive" to "very positive" and "not at all negative" to "very negative".
Experience of worst pain during delivery | 6-12 months after expected delivery
  100 mm visual analogue scale regarding the worst experience of pain during birth, using the anchors "not painful at all" and "worst pain possible".
Experience of overall pain experience during delivery | 6-12 months after expected delivery
  100 mm visual analogue scale regarding overall experience of pain during birth, again using the anchors "not painful at all" and "worst pain possible".
The Childbirth experience questionnaire | 6-12 months after expected delivery
  10 items with a 5-point Likert scale ranging from 1 (''completely disagree'') to 5 (''completely agree'') assessing the experience of childbirth, more specifically the distress and pain experienced

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Ekdahl, PhD, Principal Investigator — Depratment of Psychology, Mid Seden University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haines H, Pallant JF, Karlstrom A, Hildingsson I. Cross-cultural comparison of levels of childbirth-related fear in an Australian and Swedish sample. Midwifery. 2011 Aug;27(4):560-7. doi: 10.1016/j.midw.2010.05.004. Epub 2010 Jul 3. PMID 20598787
- [Background] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Sullivan, M.J.L., Bishop, S.R., Pivik, J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment 7: 524-532, 1995
- [Background] Carleton RN, Gosselin P, Asmundson GJ. The intolerance of uncertainty index: replication and extension with an English sample. Psychol Assess. 2010 Jun;22(2):396-406. doi: 10.1037/a0019230. PMID 20528066
- [Background] Gosselin P, Ladouceur R, Evers A, Laverdiere A, Routhier S, Tremblay-Picard M. Evaluation of intolerance of uncertainty: development and validation of a new self-report measure. J Anxiety Disord. 2008 Dec;22(8):1427-39. doi: 10.1016/j.janxdis.2008.02.005. Epub 2008 Mar 2. PMID 18395409
- [Background] Hebert, E. A., Dugas, M. J., Tulloch, T. G., & Holowka, D. W. (2014). Positive beliefs about worry: A psychometric evaluation of the Why Worry-II. Personality and Individual Differences, 56, 3-8.
- [Background] Freeston, M. H., Rhéaume, J., Letarte, H., Dugas, M. J., & Ladouceur, R. (1994). Why do people worry? Personality and Individual Differences, 17(6), 791-802. doi:10.1016/0191-8869(94)90048-5
- [Background] Sexton KA, Dugas MJ. The Cognitive Avoidance Questionnaire: validation of the English translation. J Anxiety Disord. 2008;22(3):355-70. doi: 10.1016/j.janxdis.2007.04.005. Epub 2007 Apr 25. PMID 17544253
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Van den Bussche E, Crombez G, Eccleston C, Sullivan MJ. Why women prefer epidural analgesia during childbirth: the role of beliefs about epidural analgesia and pain catastrophizing. Eur J Pain. 2007 Apr;11(3):275-82. doi: 10.1016/j.ejpain.2006.03.002. Epub 2006 Apr 18. PMID 16624602